CLINICAL TRIAL: NCT05285241
Title: Effects of Multi-direction Stepping and Weight Shifting Exercises on Balance and Gait in Stroke Patients
Brief Title: Effects of Multi-direction Stepping and Weight Shifting Exercises in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACP/OP/2016/ OL 06
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Stroke; Balance; Gait; Berg balance scale; Functional gait assessment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two arms parallel design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidirectional exercise group (Experimental): Multidirectional stepping exercises along with conventional physiotherapy were provided to the patients. Conventional physiotherapy included one-to-one range of motion exercises (10min), Strengthening exercises (10 min), Functional mat exercises (10 min), Stretching exercises (5 min), and Gait exercises (10 min).
  Interventions: Other: Multidirectional stepping exercises
- Conventional Physiotherapy Group (Active Comparator): One-to-one range of motion exercises (10min), Strengthening exercises (10 min), Functional mat exercises (10 min), Stretching exercises (5 min), and Gait exercises (10 min) were provided to the patients.
  Interventions: Other: Conventional physiotherapy group

INTERVENTIONS:
Other: Multidirectional stepping exercises — These exercises included stepping of the legs in different directions i.e. sideways, sideways and forefoot (forward), sideways and heel (backward).
  Arms: Multidirectional exercise group
Other: Conventional physiotherapy group — Conventional physiotherapy included a one-to-one range of motion exercises (10min), Strengthening exercises (10 min), Functional mat exercises (10 min), Stretching exercises (5 min), and Gait exercises (10 min)
  Arms: Conventional Physiotherapy Group

SUMMARY:
Stoke is a leading cause of disability that results not only in persistent neurological deficits but also profound physical de-conditioning that propagates stroke-related secondary disability. Several kinds of research have reported that there has been asymmetrical weight bearing on the affected side while sitting and standing resulting in impaired performance especially reaching in sitting, rising from the chair, walking, and climbing stairs. Despite the stroke patient being able to walk independently with or without the walking aids, the patient still lacks the normal movement pattern especially weight transfers on the affected side while performing such activities which subsequently decreases the patient to restrain the challenges while walking, decrease confidence in functional activities. Also, further, there hasn't been enough literature on this topic. Therefore, the objective of this study is to find out the effectiveness of multidirectional stepping and weight shifting exercises to improve dynamic balance and gait speed in stroke patients.

DETAILED DESCRIPTION:
The twenty-four subjects who fulfilled the inclusion criteria were selected for the study and were randomly assigned into two groups of 12 subjects each by simple random sampling based on inclusion criteria. First, all the subjects were assessed with a detailed neurological assessment form after the consent form was taken from the patients. The experimental group was given multidirectional stepping exercise with conventional therapy whereas are control group was given only conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke via CT Scan or MRI
* Maintain the independent standing posture for 30 sec
* Ability to walk 3 meters independently without an assistive device
* Mini-Mental status examination score >21 points
* Could communicate and understand therapist's verbal command
* Voluntary agreed to participate in the study
* Age above 18 years old
* Medically stable (e.g. recent myocardial infarction, unstable angina, ventricular tachycardia)

Exclusion Criteria:

* Visual disorders and visual deficits
* History of any neurological pathology like Parkinson's or Alzheimer's disease
* Conditions affecting balance like vertigo
* Medications affecting balance
* Dementia
* Impaired conscious level or concomitant medical illness
* Lower Motor Neuron lesions
* Anti-spasmodic medication (e.g. Baclofen, Dantrolene Sodium, etc.)
* Severe orthopedic diseases in lower extremities (e.g. Osteoarthritis, fracture, sprain, strain)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 4 weeks.
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. Minimum possible value is 0 and maximum possible value is 56. Higher score represents better outcome.
Functional gait assessment | 4 weeks.
  The Functional Gait Assessment (FGA) assesses postural stability during walking tasks in persons with gait impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No